CLINICAL TRIAL: NCT03591926
Title: A Phase 2a, 24-Week, Multi-Center, Open-Label Study Evaluating the Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of SM04646 Inhalation Solution in Subjects With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: A Study Evaluating the Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of SM04646 Inhalation Solution in Subjects With Idiopathic Pulmonary Fibrosis (IPF)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study withdrawn for business reasons prior to screening or enrolling any subjects.
Sponsor: Biosplice Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SM04646-IPF-03
Record Dates: First submitted 2018-07-09; First posted 2018-07-19 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: SM04646; IPF; nebulized; inhalation
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- "BAL" Arm (Experimental): Subjects in this arm will undergo a bronchoalveolar lavage (BAL) procedure at baseline and after two weeks of treatment.
  Interventions: Drug: SM04646
- "Non-BAL" Arm (Experimental): Subjects in this arm will not undergo any BAL procedures.
  Interventions: Drug: SM04646

INTERVENTIONS:
Drug: SM04646 — Nebulized, inhaled solution; single dose concentration dosed once per day for 12 weeks; dosing pattern will follow a 2 weeks on, 2 weeks off regimen, wherein subjects will dose 5 consecutive days of each 7 day "on" week.

SUMMARY:
SM04646-IPF-03 is a Phase 2a, multi-center, open-label study evaluating the safety and efficacy of a single inhaled, nebulized dose of SM04646 solution over a 12-week treatment regimen in subjects with mild to moderate IPF. A total of approximately 24 subjects will be enrolled in the study (approximately 12 subjects into the "non-bronchoalveolar lavage [BAL]" arm and approximately 12 subjects into the "BAL" arm). Subjects that currently do not require, have failed to tolerate, or have opted not to have treatment with pirfenidone or nintedanib will have the option of participation in the "BAL" arm or participation in the "non-BAL" arm. Subjects currently receiving treatment with pirfenidone or nintedanib must be on stable treatment for a minimum of 12 weeks prior to the Screening Visit. Subjects currently on treatment with pirfenidone or nintedanib may participate in the "non-BAL" arm only.

Eligible subjects will participate in a treatment period of 12 weeks and a follow-up period of 12 weeks. The treatment dosing pattern will follow a 2 weeks on, 2 weeks off regimen, wherein subjects will dose 5 consecutive days of each 7 day "on" week.

ELIGIBILITY:
Inclusion Criteria:

* IPF diagnosis within 5 years of study start based upon thoracic society guidelines and confirmed by Investigator at study start
* Able to walk > 150 m in 6 Minute Walk Test without the use of supplemental oxygen at study start
* Has a life expectancy of at least 12 months in the opinion of the Investigator
* Full understanding of the requirements of the study and willingness and ability to comply with all study visits and procedures
* Able to comprehend and willing to sign an informed consent form (ICF) prior to any study-related procedure being performed
* Able to tolerate and complete placebo (vehicle) inhalation for 10 minutes without experiencing a significant cough, in the opinion of the Investigator
* Subjects currently treated with pirfenidone or nintedanib must be willing to remain on their current treatment for the duration of the protocol, unless they experience rapid progression, or if, in the opinion of the Investigator, treatment adjustments are necessary

Exclusion Criteria:

* Women who are pregnant or lactating
* Women of childbearing potential who are sexually active and are not willing to use an appropriate method of birth control during the study treatment period until 90 days post study medication administration
* Males who are sexually active and not willing to use a condom, and have a partner who is capable of becoming pregnant, if neither has had surgery to become sterilized, and/or who are not willing to use an appropriate method of birth control during the study treatment period until 90 days post study medication administration
* Males unwilling to refrain from sperm donation during the study treatment period until 90 days post study medication administration
* Subjects unwilling to refrain from blood and plasma donation during the study treatment period until 90 days post study medication administration
* A history of abuse of prescription or illicit drugs within 6 months prior to study start
* Positive urine drug and alcohol screen with the exception of positive findings related to current prescription therapy at study start
* Occurrence of serious illness requiring hospitalization within 90 days prior to study start
* Presence of active infections at study start
* Current smoker or past history of smoking (e.g., cigarettes, e-cigarettes, pipes, cigars) within 6 months of study start or >50 pack years
* Use of non-inhaled tobacco- or nicotine-containing products (e.g., chewing tobacco, nicotine gum, lozenges, or patches) within 30 days prior to study start until completion of the study
* Regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for males (1 drink = 5 ounces [150 mL] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) within 30 days prior to study start until completion of the study
* Lung transplantation anticipated during the duration of the trial
* Subjects receiving treatment with pirfenidone or nintedanib that:

  1. Have been on treatment for less than 12 weeks prior to study start
  2. Have not been on a stable dose for at least 30 days prior to study start
* Subjects who are not currently on but have previously received pirfenidone or nintedanib that have not been off of pirfenidone or nintedanib for at least 30 days prior to study start
* Receipt of any of the following medication or treatment prior to study start:

  1. N-acetylcysteine prescribed for the treatment of IPF within 30 days prior to study start
  2. Previous therapeutic radiation treatment of the lungs, mediastinum, or chest wall
  3. Participation in a clinical research trial that included the receipt of an investigational product or any experimental therapeutic procedure within 30 days or 5 half-lives of the investigational product (if known), whichever is longer, prior to study start
  4. Immunosuppressive medications [e.g., methotrexate, cyclosporine, azathioprine, systemic or inhaled glucocorticosteroids with the exception of short term use of systemic glucocorticosteroids less than or equal to 10 mg of prednisone daily (or equivalent) for a non-IPF condition such as an allergic reaction or rash] within 8 weeks prior to study start
  5. Use of any therapy targeted to treat IPF (including but not limited to d-penicillamine, endothelium receptor antagonist [e.g., bosentan, ambrisentan], and interferon gamma-1B) within 30 days prior to study start
  6. Use of any cytokine modulator (etanercept, adalimumab, efalizumab, infliximab, golimumab, certolizumab, rituximab) within 90 days or 5 half-lives, whichever is longer, prior to study start
  7. A bronchodilator used within 1 week of study start
  8. SM04646
* A "bronchodilator response" at study start, defined by an absolute increase of ≥ 12% and an increase of 0.2 L in FEV1 or FVC, or both, after bronchodilator use compared with the values before bronchodilator use
* History of any of the following conditions:

  1. Pulmonary embolism or pulmonary hypertension
  2. Creatinine clearance of less than 50mL per minute
  3. Active tuberculosis (TB) infection or history of incompletely treated latent TB infection
  4. History of malignancy within the last 5 years; however, the following subjects are eligible:

     1. Subjects with prior history of in situ cancer or basal or squamous cell skin cancer that has been completely excised
     2. Subjects with other malignancies if they have been continuously disease free for at least 5 years prior to any study drug administration
     3. Subjects with prostate cancer followed by surveillance.
  5. Any connective tissue disease, including but not limited to scleroderma, systemic lupus erythematosus, rheumatoid arthritis, and polymyositis/dermatomyositis
  6. Congenital respiratory conditions (e.g., cystic fibrosis)
  7. Chronic obstructive pulmonary disease (COPD) or asthma
  8. Current or recent respiratory tract infection (e.g., pneumonia, purulent bronchitis, or viral upper respiratory tract infection) within 30 days prior to study start
  9. Acute exacerbation of IPF, in the opinion of the Investigator, within 30 days prior to study start
  10. Human immunodeficiency virus (HIV), hepatitis C, or active hepatitis B infection
  11. Clinically significant hepatic impairment (e.g., Child-Pugh A or greater severity)
  12. Symptomatic coronary artery disease, congestive heart failure (CHF) New York Heart Association (NYHA) Class II-IV, myocardial infarction (MI), or unstable angina within 6 months prior to study start
  13. Hypertension (systolic blood pressure (SBP) >160 millimeters of mercury (mmHg) or diastolic blood pressure (DBP) >100 mmHg)
  14. Hypotension (blood pressure (BP) less than 90/60 mmHg) or mean arterial blood pressure (MAP) < 65 mmHg
  15. Current use of supplemental oxygen therapy for any condition
* Subjects who are immediate family members (spouse, parent, child, or sibling; biological or legally adopted) of personnel directly affiliated with the study at the investigative site, or are directly affiliated with the study at the investigative site
* Subjects employed by Samumed Pacific Pty Ltd, or any of its affiliates or development partners (that is, an employee, temporary contract worker, or designee) responsible for the conduct of the study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 1900-01 (Estimated); Primary Completion 1900-01 (Estimated); Study Completion 1900-01 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability: treatment-emergent adverse events (TEAEs) | Week 24
  Evaluate the safety and tolerability of SM04646 as measured by TEAEs during the entire treatment period
Safety and tolerability: number of subjects with a clinically significant change from baseline in clinical laboratory tests | Week 24
  Evaluate the safety and tolerability of SM04646 as measured by the number of subjects with a clinically significant change from baseline in clinical laboratory tests
Safety and tolerability: number of subjects with a clinically significant change from baseline in vital signs | Week 24
  Evaluate the safety and tolerability of SM04646 as measured by the number of subjects with a clinically significant change from baseline in vital signs
Safety and tolerability: number of subjects with a clinically significant change from baseline in oxygen saturation | Week 24
  Evaluate the safety and tolerability of SM04646 as measured by the number of subjects with a clinically significant change from baseline in oxygen saturation
Safety and tolerability: number of subjects with a clinically significant change from baseline in electrocardiogram (ECG) parameters | Week 24
  Evaluate the safety and tolerability of SM04646 as measured by the number of subjects with a clinically significant change from baseline in ECG parameters
Plasma pharmacokinetics (PK): Cmax | Baseline and Week 10
  Measure maximum observed concentration of SM04646 (Cmax) in blood plasma
Plasma PK: tmax | Baseline and Week 10
  Measure time to SM04646 Cmax in blood plasma
Plasma PK: AUC | Baseline and Week 10
  Measure the area under the plasma concentration-time curve (AUC) for SM04646 in blood plasma
Plasma PK: t 1/2 | Baseline and Week 10
  Measure the terminal phase half-life (t 1/2) of SM04646 in blood plasma
Plasma PK: accumulation ratio | Baseline and Week 10
  Measure the accumulation ration of SM04646 in blood plasma
Change from baseline in concentration of SM04646 in BAL fluid ("BAL" arm only) | Baseline and Week 2
  Measure concentration of SM04646 in BAL fluid prior to dosing and after two weeks of dosing

SECONDARY OUTCOMES:
Change from baseline of forced vital capacity (FVC) (% predicted) | Baseline and Week 24
Change from baseline of FVC (liters) | Baseline and Week 24
Categorical analysis of FVC (% predicted) change | Baseline and Week 24
  Categories measured as "improved", "stable", "moderate decline", or "severe decline"
Time to disease progression | Week 24
  Disease progression as defined by death, absolute decline ≥ 10% in FVC (% predicted), or respiratory hospitalization
Change from baseline of forced expiratory volume in 1 second (FEV1) (% predicted) | Baseline and Week 24
Change from baseline of FEV1 (liters) | Baseline and Week 24
Change from baseline of diffusion capacity of the lung for carbon monoxide (DLCO) (% predicted corrected for hemoglobin) | Baseline and Week 24
Change from baseline of quantitative high-resolution computed tomography (HRCT) (%) and mL) | Baseline and Week 24
Change from baseline of quantitative high-resolution computed tomography (HRCT) (mL) | Baseline and Week 24
Change from baseline of qualitative HRCT | Baseline and Week 24
  Change measured as "improved", "same" or "worse"
Change from baseline of biomarker concentration isolated from serum | Baseline and Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Yazici, M.D., Study Director — Biosplice Therapeutics, Inc.
Locations (6):
- Australia (4):
  - Research Site, Camperdown, New South Wales
  - Research Site, Concord, New South Wales
  - Research Site, Bedford Park, South Australia
  - Research Site, Clayton, Victoria
- New Zealand (2):
  - Research Site, Christchurch
  - Research Site, Dunedin